CLINICAL TRIAL: NCT01467297
Title: Ceftidoren Versus Levofloxacin in the Treatment of Patients With Acute Exacerbations of Chronic Bronchitis (AECB). Multi-centre, Open-label, Randomised, Pilot Study to Evaluate the Effects of the Treatment on Serum Inflammatory Biomarkers
Brief Title: Ceftidoren Versus Levofloxacin in the Treatment of Patients With Acute Exacerbations of Chronic Bronchitis (AECB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Francesco Blasi, professor of respiratory medicine, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP1; 2011-000531-88 (EudraCT Number)
Record Dates: First submitted 2011-09-16; First posted 2011-11-08 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: COPD Exacerbation
Keywords: Chronic bronchitis; exacerbations; treatment; ceftidoren; levofloxacin; inflammation
MeSH Terms: conditions — Bronchitis, Chronic; Inflammation | interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ceftidoren (Experimental): ceftidoren 200 mg bid for 5 days
  Interventions: Drug: ceftidoren
- levofloxacin (Active Comparator): levofloxacin 500 mg once daily for 7 days
  Interventions: Drug: levofloxacin

INTERVENTIONS:
Drug: ceftidoren — ceftidoren 200 mg bid for 5 days
  Other Names: Giasion; J01D
  Arms: ceftidoren
Drug: levofloxacin — levofloxacin 500 mg once daily for 7 days
  Other Names: levoxacin; J01M
  Arms: levofloxacin

SUMMARY:
40 outpatients with exacerbations of Chronic Obstructive Pulmonary Diseases (COPD) will be enrolled in a multi-centre, open-label, randomised, pilot study. Two treatments will be compared, ceftidoren 200 mg bid for 5 days and levofloxacin 500 mg once daily for 7 days. Primary objective of the study is to evaluate the effects of the treatment on serum inflammatory biomarkers and the secondary objective is to evaluate the clinical and microbiological efficacy at the Test Of Cure visit (TOC), DAY 7-10 (end of treatment).

The study foresees 4 visits: Visit 1 (enrolment, day 1 of treatment); Visit 2 (day 2-4); Visit 3 (Test Of Cure-TOC visit, day 7-10 end of treatment), Visit 3 (Late Post Therapy assessment, Day 28-30).

The primary parameter to test the efficacy of the study medications will be the assessment of the speed of reduction of inflammatory parameters (CRP, PCT and KL6). Every reduction of 10% will be taken into account. The comparison between treatments will be performed at visit 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients with age between 40 and 75 years with no limitation of race.
2. Patients with a diagnosis of Acute Exacerbations of Chronic Bronchitis* characterized by the presence of the following three symptoms, or at least two including purulence:

   * increased dyspnoea;
   * increased of sputum volume;
   * increased of sputum purulence, that had to be confirmed macroscopically by the investigator.

     * Chronic bronchitis is characterized by cough and excessive secretion of mucus and is diagnosed when patients report production of sputum on most days over at least three consecutive months for 2 or more consecutive years (American Thoracic Society 1995).
3. FEV1 >50% of the predicted value.
4. Availability of a valid sputum specimen of broncho-pulmonary origin for microbiological evaluation obtained by either expectoration, suction, bronchoscopy or bronchial lavage. Valid samples will be characterized by < 10 squamous epithelial cells and > 25 polymorph nuclear leucocytes per low-power magnification 100x field (Wilson 2004).
5. Negative chest radiography to rule out pneumonia and active tuberculosis.
6. Written informed consent to the trial signed and dated by the patient according to the local regulations, obtained prior to all activities related to the trial.

Exclusion Criteria:

1. Hypersensitivity or allergy to antibacterial betalactams or fluoroquinolones and/or to any component of the study medications.
2. Underlying asthma.
3. Systemic corticosteroids (treatment since ≤ 2 weeks before trial drug administration) are excluded, unless patients are chronically treated (treatment for >2 weeks before trial drug administration). Corticosteroid nasal spray administration is allowed in the first 3 days of the study drug administrations only.
4. Childbearing potential where pregnancy is not excluded by pregnancy test in urine (HCG), or lactation.
5. History of tendinopathy.
6. Recent or past history of psychiatric illness or epilepsy.
7. Recent or past history of cardiac disease or rhythm disorders or clinically significant ECG abnormalities.
8. Latent or known deficiencies for the glucose-6-phosphate dehydrogenase activity.
9. Known severe hepatic and/or renal insufficiency (AST, ALT and/or creatinine levels more than twice as high as the Upper Laboratory Norm, ULN). Should laboratory data not be available when treatment is required, the patient may be conditionally enrolled.
10. Other lower respiratory tract illness: severe bronchiectasis, cystic fibrosis, or pulmonary malignancy.
11. Concurrent infections and /or neoplasm.
12. Concomitant treatment with hypoglycemic drugs.
13. Patients under treatment with fenbufen and xanthines. Patients treated with xanthines could however be recruited if plasma levels were monitored; if plasma levels exceeded concentrations of 10-15 micrograms/ml, the daily dosages of xanthines should be lowered by the Investigator (Hendels 1983);
14. Treatment with antibiotics or antibacterials within the previous week
15. Treatment with experimental drugs in the previous 4 weeks

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
serum inflammatory biomarkers | change from baseline at day 2-4 and day 7-10
  assessment of the speed of reduction of inflammatory parameters (C-reactive protein(CRP), procalcitonin( PCT) and mucin-like glycoprotein(KL6)). Every reduction of 10% will be taken into account.

SECONDARY OUTCOMES:
clinical efficacy | change from baseline to day 2-4 and day 7-10
  Clinical assessment (Vist 2 and visit 3) of signs and symptoms of acute exacerbations of Chronic bronchitis(AECB), such as sputum purulence, sputum volume, dyspnoea, cough and body temperature using a clinical score.The total scores obtained at Visit 2 and Visit 3 test of cure (TOC) will be compared with those obtained at Visit 1.
Microbiology efficacy | change from baseline to day 2-4 and day 7-10
  Microbiological assessments will be performed on valid sputum specimens At the TOC Visit, 7-10 days after the end of treatment.
  The results obtained at Visit 2 and Visit 3 test of cure(TOC) will be compared with those obtained at Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Francesco B Blasi, MD, Study Chair — University of Milan Italy
Locations (1):
- IRCCS Ospedale Maggiore Policlinico via F. Sforza 35, Milan, Italy